CLINICAL TRIAL: NCT01139606
Title: The Effect of Resistance Training With Vibrating Weights on Muscle Strength Development and Everyday Functioning of Upper Limbs in Untrained Adults
Brief Title: Vibration Training and Muscle Strength Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wingate Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0034-10-HYMC
Record Dates: First submitted 2010-06-06; First posted 2010-06-08 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Muscle Strength; Disabilities of the Arm, Shoulder and Hand

ARMS (1):
- Vibration trainig (Experimental)
  Interventions: Other: Vibration resistance training

INTERVENTIONS:
Other: Vibration resistance training — adding vibration to a standard resistance training with free-weights and checking the effect on muscle strength development and everyday functioning of upper limbs in untrained adults.

SUMMARY:
Introduction:

Vibration has been used to enhance muscle strength development during resistance training.

Aim:

To assess the effect of adding vibration to a regular resistance training program, using free weights, on muscle strength and everyday functioning of upper limbs in untrained adults

Methods:

60 healthy untrained adults, 30-65 yrs, will divide into two groups: experiment and control. Training program will include 24 sessions, over a course of 8 weeks. The experiment group will use a 1 kg vibrating weights and the control group will use a standard 1 kg free weights. Every session will include 10-15 min of 3-5 standard resistant exercises for upper limbs. Each subject will perform an Isokinetic evaluation of muscular performance, for upper limbs, in 3 occasions: before starting the program, immediately after completing the 8-weeks training program and 4 weeks afterwards, to check the chronic effect of each training regime. Each subject will complete a DASH (Disabilities of the arm, shoulder and hand) questionnaire at 4 occasions- as mentioned above and one more time, when completing the first 4 weeks of the training program, to reject any development of negative effects of the training program, such as pain or inflammation of the joints .

ELIGIBILITY:
Inclusion Criteria:

* healthy adults, ages 30-65
* not participating in resistance training for upper limbs regularly

Exclusion Criteria:

* unbalanced hypertension
* cardiovascular disfunction or disease
* pain and or/ inflammation of the neck, shoulders and arms
* pregnant women

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The effect of vibration on muscle strength development and everyday functioning during a standard resistance training for upper limbs in untrained adults. | 8 weeks of resistance training program

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Shargal, PhD, Study Director — Wingate Institute, Israel
Locations (1):
- Wingate Institute, Netanya, Israel